CLINICAL TRIAL: NCT02861521
Title: Reducing Postoperative Knee Flexion Contracture Recurrence by Correcting Leg Length Discrepancy in the Non-surgical Knee in Patients Undergoing Total Knee Arthroplasty for Primary Osteoarthritis: A Feasibility Study
Brief Title: Reducing Recurrent Knee Flexion Contracture by Correcting Leg Length Discrepancy After Total Knee Arthroplasty for OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20160109-01H; M16-16-033 (Other Grant/Funding Number: Elisabeth Bruyere Academic Medical Organizaton)
Record Dates: First submitted 2016-07-13; First posted 2016-08-10 (Estimated); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Osteoarthritis; Contracture
MeSH Terms: conditions — Osteoarthritis; Contracture

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Corrective shoe lift (Experimental): Participants will be given an external shoe lift to correct post-operative leg length discrepancy (LLD).
  Interventions: Device: Shoe lift
- Sham shoe intervention (Sham Comparator): Participants will be given a sham shoe intervention that does not correct post-operative leg length discrepancy.
  Interventions: Device: Sham

INTERVENTIONS:
Device: Shoe lift — Subjects will be given a shoe lift post-knee replacement to correct leg length discrepancy
  Arms: Corrective shoe lift
Device: Sham — Sham shoe modification
  Arms: Sham shoe intervention

SUMMARY:
Moving one's joints through their full range of motion (ROM) is crucial for health and wellbeing. Those who are unable to do so have difficulty carrying out simple activities like walking or feeding themselves. Lost joint ROM is called a contracture. Osteoarthritis (OA) is the most common form of arthritis. About a third of people with knee OA develop knee flexion contractures (KFlCs), the inability to fully straighten the knee. Having a KFlC before a knee replacement is a big risk factor for redeveloping one after the operation. Many people with a KFlC in the knee for surgery also have a KFlC in the other knee. The investigators believe that this non-surgical KFlC increases the risk of re-developing a KFlC in the surgical knee after surgery by encouraging bending of the surgical knee to avoid one leg being shorter than the other. No one has ever looked at whether fixing this leg length difference using a shoe lift would prevent this problem and there is little information to help design such a study. Here the investigators will see if testing shoe lift use for preventing KFlC is feasible. The investigators hypothesis is that a study evaluating the benefit of using a shoe lift to correct leg length difference in the non-surgical knee is feasible.

DETAILED DESCRIPTION:
Joint contractures are characterized by a restriction in the full passive range of motion (ROM) of a joint and are a major burden on public health. They restrict mobility, have a negative impact on quality of life, limit an individual's productivity and earning potential, and can prevent basic activities of daily living such as dressing and eating. The geriatric population is particularly vulnerable to contractures due to accumulated comorbidities leading to restricted joint movement and permanent loss of ROM.

A knee flexion contracture (KFlC) is a limitation in knee extension. Patients with KFlCs limp and are afflicted with a constant enhanced energy demand on the quadriceps muscle, putting them at higher risk for falls and injury. Walking is slow and abnormally tiring for those with KFlC such that patients may choose to walk less or not at all. Murphy et al. identified a significant increase in energy cost of walking with a KFlC of ≥15°. In addition, KFlCs cause a functional shortening in the affected limb resulting in a leg length discrepancy (LLD). LLDs contribute to even greater energy requirements for ambulation, worse pain due to premature joint wear, and are associated with knee osteoarthritis progression. One study identified shoe modification as a means of correcting this treatable risk factor. To the investigators' knowledge, no study has examined the effect of shoe modification on KFlC.

Contractures are associated with many conditions including arthritis. In the setting of osteoarthritis (OA), the most common arthritis and a world-leading cause of disability in the elderly, contractures are highly prevalent: over one third of 3,400 patients with OA presenting for total knee arthroplasty (TKA) had a KFlC. The burden of KFlC in OA is further compounded by the pre-operative contracture putting the patient at a higher risk for contracture, knee pain and poor outcome post-operatively. Loss of pre-operative ROM was found to be the best predictor of lost post-operative ROM.

During TKA, surgeons are often able to restore some or all knee ROM which transiently eliminates the contracture in the immediate post-operative period. Unfortunately, full ROM is lost over time in a notable proportion of patients. The overall incidence of KFlC following TKA has been reported to be between 1 to 5%. In patients with pre-operative KFlC, this has been reported as high as 15% with the resulting post-operative KFlCs still present at 3-year follow-up4. Patients who develop post-operative KFlC report less satisfaction, poorer function and more pain post-surgically. Post-operative loss of ROM has been described as one of the most common causes of readmission within the first 90 days after surgery and was identified as being the primary reason for nearly 20% of revision TKAs. These large percentages represent a significant number considering that 719,000 replacements were performed in the USA in 2010 and that the Ottawa hospital alone performs over 500 TKAs per year. KFlCs therefore contribute to increased health care costs.

Treatment of KFlC includes aggressive physiotherapy, therapeutic modalities, continuous passive ROM devices, bracing, manipulation under anesthesia, arthroscopy, open arthrolysis, or TKA revision surgery. Despite these numerous and costly options however, treatment is often unrewarding. Overall, contractures draw heavily on health care resources because of their chronic nature and poor response to treatment.

In a previous study, the investigators' group examined factors associated with KFlC in patients with end-stage OA going for TKA. By comparing those with contracture to those without, the investigators found that having a KFlC in the knee scheduled for TKA (the surgical knee) was associated with having a KFlC in the other (non-surgical) knee1. Once the surgical KFlC was corrected intra-operatively, these patients would suffer from a functionally shorter limb on the unoperated side. Given the disadvantages of walking on limbs of unequal length, patients may inadvertently flex the surgical knee when walking in order to equalize the limb lengths. By not accessing the full range of extension in the surgical knee, this could, over time, result in the re-development of a KFlC in the surgical knee. In this study the investigators propose to correct the LLD using a shoe lift for the unoperated knee with KFlC. The investigators believe this will reduce the likelihood of re-developing KFlC after TKA in the surgical knee. This simple, relatively inexpensive, intervention could reduce post-surgical morbidity, TKA revision rate and long-term costs to the healthcare system. Unfortunately, there is little data in the literature outlining the benefits of shoe lifts post-operatively.

Innovation: The investigators will use a simple inexpensive intervention (a shoe lift) to correct leg length shortening in the non-surgical limb in patients with OA and bilateral knee flexion contractures who have had a unilateral total knee replacement.

Objective: Determining the feasibility of studying the effects of shoe lift treatment on post-arthroplasty range of motion in the surgical knee in patients with bilateral pre-operative knee flexion contractures

Rationale: Post-operative KFlCs cause pain, and reduce function and patient satisfaction. They are a common cause of chronic disability and are costly and difficult to treat. Prevention of post-operative KFlC would therefore be beneficial to patients and the health care system. The investigators believe that providing a shoe lift to the non-surgical knee will reduce the incidence of developing post-operative KFlC in the surgical knee in patients with pre-operative KFlC. To the investigators knowledge, there is presently insufficient data in the literature upon which to design a study testing this hypothesis, either in terms of power analysis or outcome measures. By completing this Objective the investigators will accomplish 3 goals: (1) determine data variance for a power analysis for a future study, (2) determine if either of two validated pain and functional outcome measures are sensitive to differences in knee ROM, and (3) determine the number of subjects that the investigators are able to recruit within the timeframe of the study.

In this Objective, the investigators will recruit subjects and randomly allocate them to 1 of 2 groups, both having 1° knee OA with bilateral KFlCs who are scheduled for TKA:

Group 1: Leg length discrepancy (LLD) 2° to KFlC in the non-operated limb will be corrected using a shoe lift after TKA.

Group 2: "Sham" shoe modification that does not correct LLD in the non-surgical limb after TKA.

Hypothesis: It is feasible to design a larger randomized control trial to evaluate the pain and functional outcome benefits of using a shoe lift for the non-surgical knee post-operatively in patients with OA and bilateral pre-operative KFlCs. These benefits can be detected using a validated OA outcome tool.

During their post-operative inpatient stay, participants will have both their anatomic leg lengths measured (ASIS to medial malleolus) and will then be referred to be fitted with the appropriate shoe adjustment.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for unilateral TKA for 1° OA will be assessed for eligibility. Those meeting the American College of Rheumatology criteria for knee OA and having bilateral knee flexion contractures (KFlCs) will be recruited. KFlC will be defined as a loss of knee extension of 6 or more degrees.

Exclusion Criteria:

* Exclusion criteria include TKA for cause other than primary OA, previous septic arthritis, history of inflammatory arthritis, previous condition or known connective tissue disease that is known to affect joint range of motion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Pain assessed by visual analogue scale | Baseline (pre-op recruitment)
  Pain assessed by visual analogue scale
Pain assessed by visual analogue scale | 3 months post-knee replacement
  Pain assessed by visual analogue scale
Pain assessed by visual analogue scale | 6 months post-knee replacement
Pain assessed by visual analogue scale | 12 months post-knee replacement
Pain assessed by visual analogue scale | 24 months post-knee replacement
Pain assessed by pain subscales of Knee injury and Osteoarthritis Outcome Score (KOOS) and The Western Ontario and McMaster Universities Arthritis Index (WOMAC). | Baseline (pre-op recruitment)
  Pain assessed by pain subscales of KOOS and WOMAC.
Pain assessed by pain subscales of Knee injury and Osteoarthritis Outcome Score (KOOS) and The Western Ontario and McMaster Universities Arthritis Index (WOMAC). | 3 months post-knee replacement
  Pain assessed by pain subscales of KOOS and WOMAC.
Pain assessed by pain subscales of KOOS and WOMAC. | 6 months post-knee replacement
Pain assessed by pain subscales of KOOS and WOMAC. | 12 months post-knee replacement
Pain assessed by pain subscales of KOOS and WOMAC. | 24 months post-knee replacement
Function assessed by function subscales of KOOS and WOMAC. | 3 months post-knee replacement
  Function assessed by function subscales of KOOS and WOMAC.
Function assessed by function subscales of KOOS and WOMAC. | 6 months post-knee replacement
  Function assessed by function subscales of KOOS and WOMAC.
Function assessed by function subscales of KOOS and WOMAC. | 12 months post-knee replacement
  Function assessed by function subscales of KOOS and WOMAC.
Function assessed by function subscales of KOOS and WOMAC. | 24 months post-knee replacement
  Function assessed by function subscales of KOOS and WOMAC.

SECONDARY OUTCOMES:
Bilateral knee range of motion measured using goniometer. | Baseline (pre-op recruitment)
  Measured using goniometer
Bilateral knee range of motion measured using goniometer. | 3 months post-knee replacement
  Measured using goniometer
Bilateral knee range of motion measured using goniometer. | 6 months post-knee replacement
  Measured using goniometer
Bilateral knee range of motion measured using goniometer. | 12 months post-knee replacement
  Measured using goniometer
Bilateral knee range of motion measured using goniometer. | 24 months post-knee replacement
  Measured using goniometer
6-minute walk test | 3 months post-knee replacement
  6-minute walk test
6-minute walk test | 6 months post-knee replacement
  6-minute walk test
6-minute walk test | 12 months post-knee replacement
  6-minute walk test
6-minute walk test | 24 months post-knee replacement
  6-minute walk test
Leg length | Baseline (pre-op recruitment)
  Clinical evaluation of leg length of both lower extremities
Leg length | 3 months post-knee replacement
  Clinical evaluation of leg length of both lower extremities. Clinical leg length will be measured by a trained research assistant for both lower limbs with the patient supine, using a tape measurer from the anterior superior iliac spine to the medial malleolus with the knee maximally extended.
Leg length | 6 months post-knee replacement
  Clinical evaluation of leg length of both lower extremities. Clinical leg length will be measured by a trained research assistant for both lower limbs with the patient supine, using a tape measurer from the anterior superior iliac spine to the medial malleolus with the knee maximally extended.
Leg length | 12 months post-knee replacement
  Clinical evaluation of leg length of both lower extremities. Clinical leg length will be measured by a trained research assistant for both lower limbs with the patient supine, using a tape measurer from the anterior superior iliac spine to the medial malleolus with the knee maximally extended.
Leg length | 24 months post-knee replacement
  Clinical evaluation of leg length of both lower extremities. Clinical leg length will be measured by a trained research assistant for both lower limbs with the patient supine, using a tape measurer from the anterior superior iliac spine to the medial malleolus with the knee maximally extended.

CONTACTS AND LOCATIONS:
Overall Officials: T Mark Campbell, MD MSc FRCPC, Principal Investigator — University of Ottawa
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Data will be reported in aggregate.